CLINICAL TRIAL: NCT07223112
Title: Effectiveness of Interventions to Promote Physical Activity During Pregnancy
Acronym: SLMM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jean Davis, Associate Professor, University of Central Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 529953 clinicaltrials.gov; R03HD117025 (NIH)
Record Dates: First submitted 2025-10-15; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy; Sedentary Behavior; Insufficient Physical Activity
Keywords: Sit Less, Move More effectiveness for pregnant women; physical activity habit formation; sedentary behavior habit reversal; sedentary time disruption; wearable device; nudging; health coach; social support; behavior change
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Hybrid Model, Behavioral intervention clinical trial for effect on behavior change and implementation adaption for scale
Masking Description: Participant baseline physical activity is masked to the participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sit Less, Move More (SLMM) program intervention (Experimental): Health Coaching sessions and text messages; Fitbit sedentary time disruption, monitoring, self-regulation, exercise with a partner most days of the week to ACOG opinion 804 recommended physical activity
  Interventions: Behavioral: Sit Less, Move More (SLMM) for pregnant women

INTERVENTIONS:
Behavioral: Sit Less, Move More (SLMM) for pregnant women — Health Coach sessions and SMS texts ramp up to goal ACOG opinion 804 pregnancy physical activity; wearable device activity tracker (Fitbit) for monitoring and self-regulation, exercise with a partner for support and accountability most days of the week.

SUMMARY:
Pregnant women are more sedentary (sit, recline, lie down more) on average than non-pregnant women (more than 12 versus less than 8 waking sedentary hours/day). Sedentary behavior has been related to psychological distress, pregnancy weight gain, impaired sleep and very large size infants, while adequate physical activity has been found to improve mental health, decrease risk of high blood pressure in pregnancy and lower risk of preterm birth infants (less than 37 weeks gestation). Decreased sedentary behavior and increased physical activity may be crucial and neglected lifestyle behavior changes that can be promoted to reduce these and other maternal health and birth outcome problems among pregnant women.

DETAILED DESCRIPTION:
Interventions that decrease sedentary behavior (SB) and improve physical activity (PA) provide a path to improve maternal health and infant outcomes. Sedentary behavior (sitting, reclining, or lying while awake; activity energy expenditure of 1.5 metabolic equivalent of task [MET]) during pregnancy is a modifiable factor associated with adverse maternal health (e.g., psychological distress, gestational weight gain, impaired sleep, impaired glucose regulation, hypertension) and infant (e.g., earlier gestational age at birth, macrosomia [>4,000 grams]) health outcomes. Pregnant women are more sedentary than the average U.S. reproductive age woman (>12 hours/day vs. <8 hours/day), placing pregnant women in the highest sedentary risk category. Most pregnant women do not meet pregnancy guideline recommendations for moderate-intensity PA of 150 minutes/week. Improved PA among pregnant women is crucial to improve maternal health outcomes.

Using a behavioral clinical trial design, 60 pregnant women with singleton pregnancy (e.g., no twins) will be recruited at 8-12 weeks gestation (T1) from prenatal clinics. Participants will engage in the Sit Less, Move More (SLMM) intervention. At T1, participants complete questionnaires about SB and PA habits, weekly PA, and personal factors (e.g., demographics) and wear an ActiGraph PA tracker for 2 weeks. At Week 3, Fitbits and a SB and PA prescription will be given to participants with information on safe recommended pregnancy PA and health risks of SB while pregnant; have PA coaching (virtual 1:1 session, weekly texts); exercise with a partner at least 4 days/week; and receive Fitbit prompts for activity when SB ≥50 minutes while awake is detected. Participants also: 1) complete questionnaires at T2 (18-22 weeks) and T3 (28-32 weeks); and 2) wear a Fitbit throughout the study from Study Week 3 to 32 weeks gestation. We aim to: Aim 1) Determine the feasibility of recruitment, retention, adherence and acceptability of the SLMM intervention for pregnant women; and Aim 2) Obtain estimates of the efficacy of the SLMM intervention on daily SB, SB habit reversal, and weekly PA and PA habit for pregnant women.

The study will allow the investigators to modify SLMM, estimate its behavior change efficacy and lead to formal efficacy testing with an R01 submission to better understand pathways to improve SB and PA amongst pregnant women. This study fosters the NICHD mission to improve reproductive health and support enhanced maternal health and birth outcomes.

ELIGIBILITY:
Eligibility Criteria

* 18 to 45 years old
* speak English
* 8 to 12 weeks pregnant (gestation)
* singleton pregnancy (no twins or more)
* self-report less than 150 minutes/week of moderate-intensity physical activity
* have or are willing to identify a physical activity partner
* have a cell phone with the capacity for Fitbit application (app.); secure transmission of Fitbit data; receive coaching text messages or, if not, a computer they can use to synch the fitbit, send data, and receive email messages in lieu of texts.

Exclusion Criteria

• Women with physical activity restrictions (e.g., placenta previa) that prevent them from completing ACOG recommended pregnancy physical activity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant Females
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from first two weeks (baseline) ActiGraph device measured weekly moderate-intensity physical activity in minutes/week and time spent in sedentary behavior in hours per day | Intervention begins at 10-14 weeks gestation; 18-22 weeks gestation ActiGraph measured weekly PA & ST; 28 -32 weeks gestation ActiGraph measured weekly PA & ST; Fitbit measured weekly PA & daily ST measured 10-14 to 28-32 weeks gestation
  Change from first two weeks moderate-intensity physical activity in minutes per week and sedentary time measures in hours per day, baseline measure by participant blinded ActiGraph at 8 to 12 weeks gestation, prior to the intervention beginning with goal of pregnancy recommended moderate-intensity physical activity using CDC talk test of 150 minutes/week measured by Fitbit and sedentary time 8 hours/day or less. The intervention begins at 10 to 14 weeks gestation. ActiGraph device measured change from 8 to 12 week baseline physical activity and sedentary time as described above is measured again at 18 to 22 weeks gestation, and 28 to 32 weeks gestation in minutes of moderate-intensity physical activity per week and hours of sedentary time per day.

SECONDARY OUTCOMES:
Feasibility of recruitment for the study | 6 months (January 2026 through June 2026)
  The following metrics are used to measure this outcome:
  • Over 6 months the research team will recruit 60 participants.
Feasibility of retention in the SLMM intervention | 10 to 14 weeks gestation start of SLMM per participant through 28 to 32 weeks gestation
  The following metric is used to measure this outcome: ≥70% of participants in SLMM will be retained through 28 to 32 weeks gestation
Feasibility of adherence to the SLMM intervention | 10-14 weeks gestation through 28 to 32 weeks gestation
  ≥70% of participants in SLMM will adhere by achieving moderate-intensity physical activity ≥4 days/week as measured by Fitbit; using the Fitbit ≥10 hours/day for ≥4 days/week as measured by Fitbit; responding to ≥50% of Fitbit prompts of haptic vibration and text to move ≥4 days/week as measured by Fitbit; achieving decreased sedentary behavior by Fitbit measure by endpoint of 28 to 32 weeks gestation compared to first week of Fitbit use at 10-14 weeks gestation; complete ≥2 of 3 coach sessions as documented on coach session checklist at 10-14 weeks gestation, 18 to 19 weeks gestation and 28 to 29 weeks gestation; and receive weekly coach texts with receipt recorded in UCF text message software from 10 to 14 weeks gestation through 28 to 32 weeks gestation
Acceptability of the SLMM Intervention to participants | 18 to 22 weeks gestation and 28 to 32 weeks gestation
  ≥80% of participants in SLMM will indicate high program acceptance of all components of the intervention--coaching Fitbit use and exercise with a partner, through satisfaction items on surveys item "How satisfied are you with the SLMM program?" and open-ended question response to "How satisfied are you with the SLMM program?" following coaching sessions as recorded on coach session checklist

CONTACTS AND LOCATIONS:
Overall Officials: Jean W Davis, PhD, DNP, EdD, Principal Investigator — University of Central Florida

IPD SHARING:
Plan to Share IPD: Yes
DATA MANAGEMENT AND SHARING PLAN below and through OpenICPSR according to its terms and conditions.
  Following the study and initial publications, data will be shared per NIH - NICHD requirements. The de-identified data will be housed indefinitely in the OpenICPSR databank administered by the University of Michigan. Access occurs by open access to researchers of member organizations such as UCF and otherwise through approved requests for research purposes.
  All de-identified participant data will be stored. No PHI or identifiable participant data from this study is stored in OpenICPSR.
  Users are required to apply for access to restricted data. Additionally, non-members will be charged $825 to access the data (this includes the administrative fee to access data in the virtual data enclave) plus a $349 administrative fee for secure download." https://www.openicpsr.org/openicpsr/faqs Further details are available here: https://www.openicpsr.org/openicpsr/accessRD;jses
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared after publications and initial presentations, anticipated to be 1 year following the final data analysis 1/1/2029
Access Criteria: All de-identified participant data will be stored. No PHI or identifiable participant data from this study is stored in OpenICPSR.
  Users are required to apply for access to restricted data. Additionally, non-members will be charged $825 to access the data (this includes the administrative fee to access data in the virtual data enclave) plus a $349 administrative fee for secure download." https://www.openicpsr.org/openicpsr/faqs Further details are available here: https://www.openicpsr.org/openicpsr/accessRD;jses
URL: https://www.openicpsr.org/openicpsr/faqs